CLINICAL TRIAL: NCT04110977
Title: RAdiotherapy RElated Skin Toxicity: a Reminder App to Reduce Radiation Dermatitis Rates in Patients with Head-and-Neck Cancer
Brief Title: A Reminder App to Reduce Radiation Dermatitis Rates in Patients with Head-and-Neck Cancer
Acronym: RAREST-02
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After the planned interim analysis, the study was terminated. The start of the trial was delayed due to data protection issues and the Covid-19 pandemic. Moreover, accrual was slower than expected. Finally, funding has expired.
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Prof Dirk Rades, Chair of the Department of Radiation Oncology, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RAREST-02
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2022-12

CONDITIONS: Radiation Dermatitis; Radiation-induced Oral Mucositis
Keywords: Head-and-neck cancer; radiotherapy; radiation dermatitis; oral mucositis; reminder app
MeSH Terms: conditions — Radiodermatitis; Head and Neck Neoplasms; Stomatitis

STUDY DESIGN:
Intervention Model Description: randomized, active-controlled, parallel-group trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care supported by a Reminder App (Arm A) (Experimental): Treatment with Standard Care supported by a Reminder App, starting at the beginning of radiotherapy.
  Interventions: Device: mobile application (reminder app)
- Standard Care alone (Arm B) (Active Comparator): Treatment with Standard Care alone, starting at the beginning of radiotherapy.
  Interventions: Device: mobile application (reminder app)

INTERVENTIONS:
Device: mobile application (reminder app) — This app will remind the patients four times a day to perform skin and mouth care. Instructions are given how to properly perform skin and mouth care. The patients may postpone each required care procedure for up to 2 hours. Finally, the patients are asked to state for each procedure whether or not they performed it. To increase the patients' motivation, they will earn points for each successfully performed care procedure.

SUMMARY:
The goal of this randomized trial is to investigate whether the addition of a reminder app to standard care leads to a reduction of dermatitis and oral mucositis during radio(chemo)therapy for locally advanced squamous cell carcinoma of the head-and-neck (SCCHN). The primary endpoint is the rate of patients experiencing grade ≥2 radiation dermatitis at 60 Gy of radiotherapy. 80 patients are required per arm within the full analysis set. Taking into account that 5% of patients will not qualify for full analysis set, 168 patients should be randomized. If the addition of a reminder app to standard care will result in a significant reduction of radiation toxicity, it could become a helpful tool for these patients.

DETAILED DESCRIPTION:
The goal of this trial is to investigate whether the addition of a reminder app to standard care leads to a reduction of dermatitis and oral mucositis during radio(chemo)therapy for locally advanced squamous cell carcinoma of the head-and-neck (SCCHN).

This is a randomized, active-controlled, parallel-group trial, which will compare the following treatments of radiation dermatitis (primary endpoint) and oral mucositis in patients with SCCHN: Standard care supported by a reminder app (Arm A) vs. standard care alone (Arm B). The primary endpoint is to investigate the rate of patients experiencing grade ≥2 radiation dermatitis at 60 Gy of radiotherapy, the minimum planned total dose for all patients receiving definitive or adjuvant radiotherapy for locally advanced SCCHN with curative intention. In addition, the following endpoints will be evaluated: Radiation dermatitis grade ≥2 at the end of radiation treatment (EOT), radiation dermatitis grade ≥3 at 60 Gy and EOT, quality of life, pain, and radiation-induced oral mucositis grade ≥2 and grade ≥3 at 60 Gy and at EOT. According to sample size calculations, 80 patients are required per arm within the full analysis set. Taking into account that 5% of patients will not qualify for full analysis set, 168 patients should be randomized. The impact of the reminder app will be considered clinically relevant, if the rate of grade ≥2 radiation dermatitis can be reduced from 85% to 65%.

If the addition of a reminder app to standard care will result in a significant reduction of radiation dermatitis and oral mucositis, it could become a helpful tool for patients during radiotherapy of for SCCHN.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the head-and-neck (SCCHN)
* Indication for definitive or adjuvant radio(chemo)therapy
* Possession of and ability to use a smart phone
* Age ≥18 years
* Written informed consent
* Capacity of the patient to contract

Exclusion Criteria:

* Nasopharynx cancer
* Pregnancy, Lactation
* Treatment with epidermal growth factor receptor (EGFR)-antibodies (either given or planned)
* Expected non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Rate of radiation dermatitis grade ≥2 | until 60 Gy of radiotherapy
  at least moderate radiation-induced skin toxicity such as erythema and desquamation

SECONDARY OUTCOMES:
Rate of radiation dermatitis grade ≥2 | at the end of radiotherapy
  at least moderate radiation-induced skin toxicity such as erythema and desquamation
Rate of radiation dermatitis grade ≥3 | at 60 Gy of radiotherapy and at the end of radiotherapy
  severe radiation-induced skin toxicity such as erythema and desquamation
Pain score | prior to radiotherapy, weekly during radiotherapy, at 60 Gy and at the end of radiotherapy
  Pain within the radiation fields measured with a self-rating analogue scale ranging from 0 (no pain) to 10 (maximum pain) points; higher values represent worse outcomes.
Rate of radiation-induced oral mucositis grade ≥2 | at 60 Gy of radiotherapy and at the end of radiotherapy
  at least moderate radiation-induced inflammation of the oral mucosa
Rate of radiation-induced oral mucositis grade ≥3 | at 60 Gy of radiotherapy and at the end of radiotherapy
  severe radiation-induced inflammation of the oral mucosa

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Rades, Professor, Principal Investigator — Dept. of Radiation Oncology, University of Lübeck, Germany
Locations (4):
- Germany (2):
  - Medical Practice for Radiotherapy and Radiation Oncology, Hanover, Lower Saxony
  - Dept. of Radiation Oncology, University of Lübeck, Lübeck, Schleswig-Holstein
- Spain (2):
  - Dept. of Radiation Oncology, Hospital Universitario y Politecnico La Fe,, Valencia, Valencia
  - Department of Radiation Oncology, Cruces University Hospital/ Biocruces Health Research Institute, Barakaldo, Vizcaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rades D, Narvaez CA, Doemer C, Janssen S, Olbrich D, Tvilsted S, Conde-Moreno AJ, Cacicedo J. Radiotherapy-related skin toxicity (RAREST-02): A randomized trial testing the effect of a mobile application reminding head-and-neck cancer patients to perform skin care (reminder app) on radiation dermatitis. Trials. 2020 May 25;21(1):424. doi: 10.1186/s13063-020-04307-0. PMID 32450921